CLINICAL TRIAL: NCT07126392
Title: You and Me Healthy: Test to Treat
Acronym: YMTT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00112479; 1U01MD018294-01 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: COVID - 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic dramatically increased health disparities. In the United States, >79 million have been infected with SARS-CoV-2 and >900,000 died, but cases and deaths disproportionately affect underserved populations. Novel treatments early in disease may transform the pandemic's course, but strategies that address disparities in timely testing and treatment access are essential to maximize impact. To address profound COVID-19 disparities, testing strategies should be developed together with community-trusted organizations in high-need areas identified with risk assessment strategies to address barriers to test access, determine infrastructure needs, and position testing to promote timely access, awareness and education, and engagement with health systems and local resources. The You & Me Healthy (YMH) Toolkit is a guide to develop academic-community partnerships in underserved communities in response to public health threats. In this application, the investigators will evaluate the toolkit's role in preparing community-based test distribution and test and treat responses to the next phase of the COVID-19 pandemic in underserved populations.

Widening COVID-19 health and education disparities will have a profound impact for generations, with infections and deaths disproportionally affecting underserved populations that have been historically marginalized. Inequitable risk of COVID-19 infection and unequal access to care have been observed among lower socio-economic and racial/ethnic minorities with higher hospitalization rates, lower recovery rates, and higher mortality. As outlined at the core of Public Health 3.0, local communities will lead the charge in taking public health to the next level and ensure its continued success. Within this framework community members serve as partners for research, and both community and research resources are leveraged to address social, environmental, and economic conditions that magnify health disparities in communities. Community engagement is increasingly being recognized as enhancing research quality and relevance to public health practice. Benefits of engaging communities have been reported in all stages of research including 1) identifying key research questions based on firsthand knowledge and insight from the field; 2) designing informed consent processes and research protocols that meet the needs of the community; 3) adapting public health interventions to be context-relevant; 4) identifying implementation processes to promote public health intervention feasibility and adoption; and 5) disseminating research results to make information more accessible.

DETAILED DESCRIPTION:
This observational study is a direct-to-participant study that distributes at-home, self-administered, COVID-19 testing kits to people in designated communities. The investigators are working together with two anchor partners (Merced County United Way and Pitt County Health Department), who will coordinate directly with 10 local partners each to distribute 10,000 COVID test kits each (20,000 tests) at community-based testing events (location and timing based on community partner guidance) over a 15-month period. All eligible and consented participants at testing events will complete basic data collection including demographics, COVID-19 questions, additional testing satisfaction survey questions and contact information using the Colectiv. Community partners will also complete community partner engagement surveys using the app. Participants will also receive guidance on COVID-19 mitigation, health-promoting resource linkage, and accessible/affordable therapeutics if they test positive for COVID-19.

This proposal will evaluate a systematic and scalable community-engaged test and treat protocol that provides rapid access to COVID-19 at-home tests for self-administration, "next steps" guidance and education, and information on local resources to facilitate treatment in underserved populations. The protocol will be designed and implemented in two communities, Pitt County, NC, and Merced County, CA, in collaboration with key community partners over a 15-month period. As part of this test and treat protocol, the investigators will evaluate a community engagement toolkit, the You & Me Healthy (YMH) Toolkit, as a resource to implement community-based test distribution and test and treat responses in underserved populations. The central hypothesis is that the YMH Toolkit will enable rapid design and implementation of a community driven, scientifically robust, and impactful COVID-19 test and public health intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported primary residence within the pre-identified communities
* Age≥ 8 years at enrollment
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Under 8 years old
* Resides outside of pre-identified communities

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This observational study is a direct-to-participant study that distributes at-home, self-administered, COVID-19 testing kits to people in designated communities. The investigators are working together with two anchor partners (Merced County United Way and Pitt County Health Department), who will coordinate directly with 10 local partners each to distribute 10,000 COVID test kits each (20,000 tests) at community-based testing events (location and timing based on community partner guidance) over a 15-month period.
Sampling Method: Non-Probability Sample
Enrollment: 913 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Number of consented participants | Baseline
  Participants completed the informed consent
Total number of home test kits distributed. | Up to 2 years
  Participants received home test kits that were distributed at various events and locations
Proportion of at-home test results that were reported | Baseline; 3 days
  Participants completed a survey regarding the reporting of results.
Proportion of positive test participants receiving information on COVID-19 next steps. | 1 hour of reporting positive results
  Participant received an email that detailed local services.
Proportion of participants with positive test results who receive a link to a community testing site | 1 hour of reporting results
  Participants received an email with information on local testing sites
Proportion of positive test participants who are provided a link to treatment | 1 hour of reporting results
  Participants were sent an email that included local treatment options.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M D'Agostino, DPH, MS, MEd, MA, Principal Investigator — Duke Clinical Research Institute
Locations (2):
- United States (2):
  - United Way of Merced California, Merced, California
  - Pitt County Health Department, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No